CLINICAL TRIAL: NCT06128174
Title: Pulsed Field Ablation for Long-Standing Persistent Atrial Fibrillation (LS-PersAFone)
Brief Title: LS-PersAFone: Pulsed Field Ablation for Long-Standing Persistent Atrial Fibrillation
Acronym: LS-PersAFone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivek Reddy (Other)
Responsible Party: Sponsor-Investigator, Vivek Reddy, EP Division Director, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-23-01039
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Long-standing Persistent AF
Keywords: Long-standing Persistent AF; Persistent Afib greater than 1 year; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Prospective Multicenter Single-Arm Investigator-Initiated IDE study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients with longstanding persistent atrial fibrillation (AF) (Experimental): All subjects will undergo Pulmonary vein isolation (PVI) and Posterior wall isolation (PWI) with the Farapulse catheter.
  Interventions: Device: Farawave PFA catheter

INTERVENTIONS:
Device: Farawave PFA catheter — The FARAWAVE Pulsed Field Ablation Catheter (FARAWAVE Catheter) is a flexible tube with electrodes at the end, which is inserted through a blood vessel in your groin. The study doctor will use the FARAWAVE Catheter to deliver the pulsed electrical energy to ablate (destroy) the heart tissue. This process is designed to create a scar in the heart tissue, stopping the unwanted electrical signals that cause the atrial fibrillation.

SUMMARY:
This is a prospective, single-arm trial. The objective of the study is to determine the rate of atrial arrhythmia recurrence after pulmonary vein isolation (PVI) plus posterior wall isolation (PWI) using the Farawave PFA catheter in patients with longstanding persistent atrial fibrillation (AF). The trial will be conducted at as many as 10 US sites. Upon completion of site initiation, enrollment is expected to accrue at a rate of 10 patients per month. Total enrollment is expected to consist of 100 subjects. Accrual is expected to take 18 months, and all patients will be followed for 12 months post randomization.

This study will be completed in 2 phases. There will be a 20 subject pilot phase, enrolled at one site (Mount Sinai). After completion of the pilot phase, the FDA will be provided with acute safety data (1 month). During the FDA's review of the pilot phase, enrollment may continue at the initial site. Also, IRB submissions at other prospective sites (up to a total of 10) may be initiated. Upon receipt of the go-ahead from FDA and after consultation with the study sponsor, the second phase of the study (to enroll 100 total subjects) will be performed. This research study currently has approval to enroll 25 patents. Should FDA grant approval to continue the study, the research team will expand as above and update this posting.

DETAILED DESCRIPTION:
Among patients with paroxysmal AF, numerous randomized studies have demonstrated the efficacy of catheter ablation as compared with anti-arrhythmic therapy to prevent arrhythmia recurrence. However, among patients with long-standing persistent AF the efficacy of catheter ablation remains particularly poor, with long-term freedom from Atrial Tachycardia AT/AF off anti-arrhythmic medications generally as low as 30% after one procedure. Multiple catheter ablation procedures are usually required in long-standing persistent AF to achieve arrhythmia suppression.

Although pulmonary vein isolation (PVI) has been the main focus of catheter ablation for atrial fibrillation, as a lesion set it is insufficient for long-standing persistent AF. Electrical isolation of the posterior wall has been proposed as an adjunctive lesion set to PVI for patients with persistent and long-standing persistent AF. The left atrial posterior wall has a common embryological origin with the pulmonary veins, and differences in fiber orientation at the intersection of the pulmonary veins and the LA posterior wall may contribute to localized re-entrant circuits and subsequent AF. In addition, the posterior wall is a site of parasympathetic innervation that could act as a non-pulmonary vein trigger for AF. Typically, posterior wall isolation (PWI) during catheter ablation involves the creation of lines between the superior edge of the left- and right-sided PVI lesion sets, as well as between the inferior edges of the left- and right-sided lesion sets. Another approach involves the delivery of lesions throughout the posterior wall to target any electrical activity.

Observational studies of PWI have suggested that it improves outcomes over PVI in persistent AF. However, randomized trials of catheter ablation for PWI have not shown clinical benefit over PVI. An important possible reason for the negative results of the randomized trials is the difficulty achieving durable PWI. In fact, a recent clinical trial of a hybrid epicardial/endocardial ablation to achieve PVI and PWI was compared with a standard endocardial catheter ablation set of PVI and a roof line. The CONVERGE clinical trial of 153 patients with persistent and long-standing persistent AF showed significantly higher rate of AF burden reduction in the treatment group (74% versus 55%) by 18 months. The durability of PWI through epicardial ablation may be a major reason for the increased efficacy in the hybrid ablation group.

Left atrial posterior wall ablation is also supported by 2 important mechanistic studies-1 surgical (HISTORIC-AF) and 1 catheter based (PersAFone). Like in CONVERGE, HISTORIC-AF evaluated a 2-procedure strategy of a minimally invasive, thoracoscopic epicardial RF tool to create a posterior box lesion isolating all PVs and the posterior wall en bloc; followed 1 month later by catheter-based endocardial touch-up ablation of residual conduction gaps. This multicenter, prospective, nonrandomized study of 100 patients (32% with PerAF, 68% with longstanding PerAF) used implantable loop recorders (ILRs) for continuous ECG monitoring for AF recurrence, and nonetheless demonstrated an excellent 1-year maintenance of sinus rhythm rate of 88%. In PersAFone, patients with PerAF underwent PVI + PWI using the Farawave pulsed field ablation (PFA) catheter. While this trial only included 25 patients, the trial was notable for a design which included remapping at 3 months (demonstrating durable PWI in all patients) with any necessary touch-up ablation performed. Following this, the one-year freedom from AF recurrence was 92±5.4%.

PFA for AF offers very promising efficacy for PVI, with ~96% durability of isolated veins at 90-day remapping. Furthermore, studies of PFA for PVI have also shown an extremely low risk of esophageal injury.

Together, these data support a PFA-based PVI+PWI strategy as a simple, safe, fast approach to treat this troublesome population of long-standing PerAF patients. Accordingly, the research team proposes a prospective study of PVI and PWI for patients with longstanding PerAF, using PFA in order to minimize the risk of esophageal injury and maximize the likelihood of durable catheter-based ablation lesions. The research team seeks to obtain precise estimates of arrhythmia recurrence post-ablation through ILRs in follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Long-standing Persistent AF (>1 year continuous AF)
* Planned for a first-ever AF ablation procedure
* Left ventricular ejection fraction >30% (as assessed within 6 months of randomization)

Exclusion Criteria:

* Prior left atrial ablation or left atrial surgery (including mitral valve surgery)
* Hypertrophic cardiomyopathy
* Major cardiac surgery within 6 months preceding the consent date
* Within 3 months preceding the consent date:

  * Stroke, TIA, intracranial bleeding
  * Any thromboembolic event
  * Carotid stenting or endarterectomy
* Life expectancy less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with freedom from recurrent atrial arrhythmias | post 3 month blanking period till end of study at 12 months
  Number of participants with freedom from recurrent atrial arrhythmias (AF/AT/AFL) (post 3-month blanking), assessed as time to first recurrence. AF/AT/AFL will be defined as an episode of the corresponding arrhythmia that is recorded for review, where the recording contains at least 30 seconds of continuous interpretable signal. An exception is a 12-lead ECG where the arrhythmia occurs during the entire tracing and the continuous interpretable signal is 10 seconds or longer.

SECONDARY OUTCOMES:
Proportion with post-blanking period AF burden <12% by device interrogation | end of study at 12 months
  Proportion with post-blanking period AF burden <12% by device interrogation. The overall burden of AF will be assessed in the treatment and control groups, and the proportion of patients in each group with AF burden <12% will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine; William Whang, MD, Principal Investigator — Icahn School of Medicine
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data not available/not applicable.